CLINICAL TRIAL: NCT05026424
Title: Glucose and Insulin Response in Adults with Type 2 Diabetes
Brief Title: Glycemic Response in Adults with Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21.04.US.HCN
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This will be a randomized crossover design. The subjects will be randomized to one of two interventions on two separate study days, one week apart.
Who Masked: Participant
Masking Description: Site pharmacy will not be blinded to product assignment, study staff and participants will be blinded to product assignment. Product will be provided in unlabeled cups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: Oral Nutrition Supplement Control (Placebo Comparator): The control study intervention is an oral drink that contain protein, carbohydrate and fat and are intended for use as supplemental nutrition.
  Interventions: Other: Balance oral nutritional drink - control
- Active Comparator: Oral Nutrition Supplement Test (Active Comparator): The test study intervention is an oral drink that contain protein, carbohydrate and fat and are intended for use as supplemental nutrition for people living with diabetes.
  Interventions: Other: Balance oral nutritional drink - test

INTERVENTIONS:
Other: Balance oral nutritional drink - control — Drink 1 cup of liquid nutrition product that contains protein, carbohydrate and fat intended for use as supplemental nutrition.
  Arms: Active Comparator: Oral Nutrition Supplement Control
Other: Balance oral nutritional drink - test — Drink 1 cup of liquid nutrition product that contains protein, carbohydrate and fat designed for people living with diabetes and intended for use as supplemental nutrition.
  Arms: Active Comparator: Oral Nutrition Supplement Test

SUMMARY:
This will be a randomized crossover design with oral nutrition supplement interventions.

DETAILED DESCRIPTION:
This will be a randomized crossover design with two oral nutrition supplement interventions. The subjects will be randomized to one of two interventions on two separate study days, one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years
* Type 2 diabetes controlled with diet or diet and metformin (Glucophage)
* Hemoglobin A1C less than 9.0%
* Fasting blood glucose less than 180 mg/dl
* Hematocrit levels within normal limits
* Having obtained his/her informed consent

Exclusion Criteria:

* Abnormal thyroid function
* Creatinine >2.0 mg/dl
* Potassium <3.5 mEq/l
* Gastrointestinal disease: ulcer, gastritis, diarrhea, gastroparesis, vomiting
* Currently unstable diabetes or under treatment for cancer, heart disease, renal disease
* Patients with anemia
* Current insulin therapy or insulin therapy within the past month
* Patient who are pregnant
* Allergies to milk, soy or any component of the test product
* Patient who in the investigators assessment cannot be expected to comply with treatment
* Patients with anemia
* Currently participating in another clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Post-prandial glycemic markers | [Time Frame: Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes]
  Area under the blood glucose curve (AUC 0-240 minutes)

SECONDARY OUTCOMES:
Post-prandial insulin markers | [Time Frame: Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes]
  Area under the insulin curve (AUC 0-240 minutes)
Insulinogenic index | [Time Frame: Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes]
  Insulinogenic index (change in Ins30/change in Glu30)

CONTACTS AND LOCATIONS:
Overall Officials: Krysmaru Araujo Torres, MD, Study Director — Nestle Health Science
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No